CLINICAL TRIAL: NCT02979886
Title: Effects of Single Nucleotide Polymorphism of GnRH Receptor Genes on Clinical Response to Pituitary Down Regulation in IVF Patients
Brief Title: Effects of SNP of GnRH Receptor Genes in IVF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Miao benyu (Other)
Responsible Party: Sponsor-Investigator, Miao benyu, the associated professor, First Affiliated Hospital of Zhongshan Medical University
Organization: First Affiliated Hospital of Zhongshan Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FirstZhongshanMU
Record Dates: First submitted 2016-11-27; First posted 2016-12-02 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Infertility, Female
Keywords: single nucleotide polymorphism,GnRH receptor, IVF
MeSH Terms: conditions — Infertility, Female | interventions — ricin A-GnRH conjugate; Triptorelin Pamoate; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- triptorelin (Experimental): GnRH-a will be given everyday to the patient undergoing IVF treatment from middle luteal phase to the day of HCG. After 14 days of injection, serum FSH/LH/E2 will be checked. Then ovarian stimulation will be started by giving daily subcutaneous injection of recombinant FSH 150~300 IU. An appropriate dose of HMG (75~150 IU) will be added when follicles are larger than 12~14mm in diameter. When one leading follicle is >18mm in diameter, or two follicles are >17mm in diameter, or three follicles are >16mm in diameter, final ovulation will be triggered by a single injection of HCG 4,000~10,000 IU or Ovidrel® 250μg (equivalent to HCG 6,500 IU)
  Interventions: Drug: GnRH-a; Drug: Human Menopausal Gonadotropins

INTERVENTIONS:
Drug: GnRH-a — the hormone reaction to the down regulation of the patients
  Other Names: triptorelin
Drug: Human Menopausal Gonadotropins — the effects on the serum LH level of day of HCG
  Other Names: menopur

SUMMARY:
Gonadotropin-releasing hormone analogue (GnRH-a) "long protocol" is a protocol for pituitary down-regulation in IVF. However, it is common in clinic that some patients are hypersensitive to pituitary down-regulation and have pituitary oversuppression, resulting in prolonged ovarian stimulation and increased consumption of exogenous gonadotropin(Gn). On the other hand, some patients may have insufficient pituitary down-regulation, which can affect the synchronization of ovarian follicles and consequently reduce the number of oocytes retrievable and lower the pregnancy rate. The differences in responses to GnRH-a among patients may be associated with the SNP of their GnRH receptor genes. It has been reported that mutations in GnRH receptor genes could change their binding affinity to the ligands, thus affecting the outcome of pituitary down-regulation. So far 20 non-synonymous mutations on the GnRH receptor genes have been reported, which can affect the function of GnRH receptor and are highly associated with disorders such as endometriosis and sexual precocity. However, the correlation between the SNP of GnRH receptor genes and the outcome of pituitary down-regulation in IVF has not been reported.

The purpose of this study is to analyze the correlation between single nucleotide polymorphism (SNP) of GnRH receptor genes in infertile female patients and the extent of pituitary down-regulation by short-acting GnRH-a long protocol, with the goal to achieve individual down-regulation protocols based on the patients' SNP haplotypes of GnRH receptor genes and to improve the success rate of assisted reproductive technology.

DETAILED DESCRIPTION:
Short-acting GnRH-a will be administered daily since the mid-luteal phase for pituitary down-regulation. 14 days after down-regulation,serum levels of follicle stimulating hormone (FSH), luteinizing hormone (LH) and E2 will be measured. Meanwhile, about 2ml of peripheral blood will be preserved for SNP analysis of the GnRH receptor genes. Once the patients are judged to achieve pituitary down-regulation, ovarian stimulation will be started. B-mode ultrasonography and determination of hormone levels will be performed regularly according to the course of follicle maturation. An appropriate dose of human menopause gonadotropin (HMG) (75~150IU) will be added when follicles are larger than 12~14mm in diameter. When one leading follicle is >18mm in diameter, or two follicles are >17mm in diameter, or three follicles are >16mm in diameter, final ovulation will be triggered by a single injection of human chorionic gonadotropin (HCG) 4,000~10,000 IU or Ovidrel® 250μg (equivalent to HCG 6,500IU).Oocyte retrieval guided by vaginal ultrasonography will be conducted 35~36 hours after HCG or Ovidrel®injection.Fertilization and embryo culture will be performed according to the standard IVF or intracytoplasmic sperm injection (ICSI) protocol.Embryo transfer and cryopreservation will be performed 3~5 days after oocyte retrieval. Luteal support will be provided after embryo transfer according to the Center's routine practice. Serum β-HCG level will be measured 12~14 days after embryo transfer to determine biochemical pregnancy, and transvaginal ultrasonography will be performed 4~5 weeks after embryo transfer to determine clinical pregnancy.

For data analysis, patients will be divided into two groups according to their serum LH level on day 14 after pituitary down-regulation - one group of patients with an LH level above the median of the group and another group of patients with an LH level below the median of the group.Comparisons will be made between the two groups in the following aspects: 1) age; BMI; basal levels of LH, FSH and prolactin (PRL); serum levels of FSH, LH, E2 and progesterone on the day of HCG injection; the numbers of oocytes retrieved, the number of cleavage, the number of transferrable embryos, the number of embryos transferred and the clinical pregnancy rate; and 2) genotyping results at the 11 SNP loci of the GnRH receptor genes.

ELIGIBILITY:
Inclusion Criteria:

* regular periods of spontaneous menstruation (23~35 days)
* basal serum FSH <12 IU/L
* use of short-acting GnRH-a long protocol for pituitary down-regulation.

Exclusion Criteria:

* polycystic ovary syndrome (PCOS)
* hypothalamic-pituitary lesions
* use of oral contraceptives
* treated with a GnRH-a within 3 months before the start of GnRH-a treatment for this study
* failure to sign informed consent form.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the evidence of the correlation between single nucleotide polymorphism (SNP) of GnRH receptor genes in infertile female patients and the extent of pituitary down-regulation by short-acting GnRH-a long protocol | two years

CONTACTS AND LOCATIONS:
Overall Officials: benyu miao, Study Director — the first affiliated hosptial of zhongshan university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noel SD, Kaiser UB. G protein-coupled receptors involved in GnRH regulation: molecular insights from human disease. Mol Cell Endocrinol. 2011 Oct 22;346(1-2):91-101. doi: 10.1016/j.mce.2011.06.022. Epub 2011 Jun 29. PMID 21736917
- [Result] Valkenburg O, Uitterlinden AG, Piersma D, Hofman A, Themmen AP, de Jong FH, Fauser BC, Laven JS. Genetic polymorphisms of GnRH and gonadotrophic hormone receptors affect the phenotype of polycystic ovary syndrome. Hum Reprod. 2009 Aug;24(8):2014-22. doi: 10.1093/humrep/dep113. Epub 2009 Apr 29. PMID 19403562
- [Result] Caronia LM, Martin C, Welt CK, Sykiotis GP, Quinton R, Thambundit A, Avbelj M, Dhruvakumar S, Plummer L, Hughes VA, Seminara SB, Boepple PA, Sidis Y, Crowley WF Jr, Martin KA, Hall JE, Pitteloud N. A genetic basis for functional hypothalamic amenorrhea. N Engl J Med. 2011 Jan 20;364(3):215-25. doi: 10.1056/NEJMoa0911064. PMID 21247312